CLINICAL TRIAL: NCT06466434
Title: Prebiotic Food-enriched Diet (PreFED) to Enhance the Microbiome and Response to First-line Immunotherapy in Unresectable Melanoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2024-0387; NCI-2024-05150 (Other: NCI-CTRP Clinical Registry)
Record Dates: First submitted 2024-06-14; First posted 2024-06-20 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Unresectable Melanoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Prebiotic food-enriched diet (PreFED) (Experimental): Participants will receive prebiotic food-enriched snacks and supportive nutritional counseling to increase prebiotic foods in the diet.
  Interventions: Other: Prebiotic Food-Enriched Diet

INTERVENTIONS:
Other: Prebiotic Food-Enriched Diet — Given by PO

SUMMARY:
To learn about the possible effects of a prebiotic food-enriched diet (PreFED) targeting the gut microbiome in participants with melanoma who are starting immune checkpoint blockade (ICB) therapy.

DETAILED DESCRIPTION:
Primary Objectives

• Evaluate the effect of dietary intervention on the abundance of Faecalibacterium in stool samples from baseline to 12 weeks

Secondary Objectives

* Determine the best overall response rate (BORR) to PreFED + ICB regimens and landmark ORR at 12 weeks (intervention) and 24 weeks (maintenance)
* Determine progression-free survival (PFS) and overall survival (OS) with PreFED + ICB regimens
* Compliance and adherence to the dietary intervention at 12 weeks and maintenance at 24 weeks
* Determine the safety (diet-related AEs) and tolerability (GSRS-IBS) of the dietary intervention at 12 weeks and maintenance at 24 weeks
* Assess the rate of immune related adverse events in patients on ICB regimens receiving dietary intervention at 12 weeks and maintenance at 24 weeks
* Assess the effects of dietary intervention on systemic and tumor immunity
* Assess the effect of dietary intervention on overall gut microbiome composition and networks at 12 weeks and maintenance at 24 weeks
* Assess the effects of dietary intervention on gut metabolic output and systemic metabolism at 12 weeks and maintenance at 24 weeks
* Assess the effects of dietary interventions on quality of life and other patient reported outcomes (PROs) at 12 weeks and maintenance at 24 weeks

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years old
* English-speaking
* Body mass index (BMI) 18.5-45 kg/m2
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically confirmed stage III/IV, unresectable cutaneous, uveal, acral or mucosal melanoma. Asymptomatic brain metastases are allowed.
* Planned initiation of 1st line standard-of-care approved immune checkpoint blockade (anti-PD1 +/- anti-CTLA4 or anti-LAG3 inhibitors) in the metastatic setting (prior ICB in the adjuvant setting is allowed.
* Returning to MD Anderson for restaging and follow-up (ICB treatment may occur locally)
* Measurable disease per RECIST 1.1 or RANO criteria. Up to 10 patients without measurable can be enrolled.
* WOCP must have negative UPT within 1 week of beginning dietary intervention.
* Self-reported willingness to eat the provided foods (with some tailoring to their food preferences)
* Self-reported willingness to comply with scheduled visits, undergo venipuncture, provide stool samples.

Exclusion Criteria:

* Previous ICB treatment in the metastatic setting
* History of inflammatory bowel disease, total colectomy, or bariatric surgery.
* Currently taking steroids > Prednisone 10 mg/day or equivalent
* Medical contraindications to the Intervention Diet as determined by the treating physician.
* Self-reported major dietary restrictions, including but not limited to relevant food allergies, celiac disease, or diets such as vegan, ketogenic, extended fasting.
* Insulin-dependent diabetes or condition requiring bile acid sequestrants
* Unable or unwilling to undergo study procedures.
* IV antibiotic use in the past month or oral antibiotic use in past 2 weeks.
* Regularly taking supplements containing prebiotics, fiber and/or probiotics, and unable/unwilling to discontinue for the purpose of the study.
* Current smoker or heavy drinker (defined as >14 drinks per week) or current illicit drug use.
* Currently pregnant, planning to become pregnant, or lactating.
* Concurrent malignancy requiring systemic therapy other than hormonal therapy.
* Cognitively impaired adults

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2027-06-30 (Estimated); Study Completion 2029-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the effect of dietary intervention on the abundance of Faecalibacterium in stool samples from baseline. | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Erez Baruch, MD,PHD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org